CLINICAL TRIAL: NCT00298311
Title: An RCT to Evaluate the Effect of Home-Based Peer Support on Maternal-Infant Interaction, Infant Health Outcomes, and Postpartum Depression
Brief Title: Effect of Home-Based Peer Support on Maternal-Infant Interaction and Postpartum Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Research Institute for Social Policy (Other)
Collaborators: Women's Health Research Unit (Unknown); Social Support Research Program (Unknown); University Health Network, Toronto (Other); Edmonton Mental Health Services (Unknown); Canadian Mental Health Association (Other); Pediatric Rehabilitation Services (Unknown); Department of Health and Wellness, NB (Unknown)
Responsible Party: Principal Investigator, Dr. Nicole LeTourneau, Professor, University of Calgary
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Health Services Research
Other Study IDs: PPD MOD
Record Dates: First submitted 2006-03-01; First posted 2006-03-02 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- mci guidance & peer social support (Experimental): home visits to promote maternal-child interaction & social support
  Interventions: Behavioral: mci guidance peer support
- peer social support (Sham Comparator): social support
  Interventions: Behavioral: mci guidance peer support

INTERVENTIONS:
Behavioral: mci guidance peer support — 12 weeks of home visits by peer mentor recovered from PPD and Keys to Caregiving (NCAST, 1990) program

SUMMARY:
The objective of this study is to examine the impact of a home-based peer support intervention for mothers affected by postpartum depression (PPD) and for their infants.

DETAILED DESCRIPTION:
This controlled study will help establish the link between support for maternal caregiving, maternal-infant interaction, infant neuroendocrinology and infant cognitive and social development. The primary hypothesis predicts that home-based peer support will improve maternal-infant interactions. Secondary hypotheses predict that home-based peer support will: improve infants' cognitive development; improve infants' social development; decrease average daily salivary cortisol levels in infants; reduce maternal depressive symptomatology; and improve maternal perceptions of social support.

ELIGIBILITY:
Inclusion Criteria:

* Eligible mothers will be identified as experiencing symptoms of PPD and scores >12 on the Edinburgh Postnatal Depression Scale.
* Mothers must speak English or French.
* Mothers will not be excluded for taking anti-depressant or anti-psychotic medication, using other interventions for PPD, or reporting a history of mental illness;
* The infant must be full-term, in the care of the mother and between 3 to 6 months of age at initial enrollment.

Exclusion Criteria:

* Infants who have been admitted to the NICU
* Infants will be excluded if medicated with corticosteroids

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-11; Primary Completion 2009-02 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
maternal-infant interaction | 12 months

SECONDARY OUTCOMES:
cognitive development | 12 months
social development | 12 months
salivary cortisol | 12 months
depressive symptomatology | 12 months
social support | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Letourneau, PhD, Principal Investigator — University of Calgary

REFERENCES:
- [Derived] Yonemoto N, Nagai S, Mori R. Schedules for home visits in the early postpartum period. Cochrane Database Syst Rev. 2021 Jul 21;7(7):CD009326. doi: 10.1002/14651858.CD009326.pub4. PMID 34286512